CLINICAL TRIAL: NCT05728788
Title: Correlation Between Early Myocardial Injury and Intestinal Flora Changes Associated With Oncology Drug Therapy
Brief Title: Correlation Between Myocardial Injury and Intestinal Flora Changes Associated With Oncology Drug Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021598
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Cancer Therapy-related Cardiovascular Toxicity
MeSH Terms: interventions — Antineoplastic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will test the collected fecal samples for 16S-rDNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with antineoplastic agents: 50 patients treated with antineoplastic agents will be enrolled.
  Interventions: Drug: Antitumor drugs

INTERVENTIONS:
Drug: Antitumor drugs — Anthracyclines, immune checkpoint inhibitors, monoclonal antibodies, and tyrosine kinase inhibitors

SUMMARY:
The purpose of this study was to explore the relationship between early myocardial injury caused by tumor drug therapy and intestinal microbial structure changes by echocardiographic two-dimensional speckle tracking technique and intestinal microflora structure detection.

DETAILED DESCRIPTION:
This is a monocentric prospective cohort study in which 50 patients treated for malignant tumors will be included. All participants will be followed for 6 months after the initiation of oncology drug therapy. Echocardiography and 2D speckle tracking will be performed and stool and blood samples will be tested before treatment initiation and at 3 and 6 months after initiation.

ELIGIBILITY:
Inclusion Criteria:

* With malignant tumors
* Will receive antitumor drugs
* Could receive regular follow-up for 6 months
* Written informed consent

Exclusion Criteria:

* Satisfactory echocardiographic images could not be obtained
* Cardiomyopathy
* Coronary artery disease
* Heart failure
* Arrhythmia requiring intervention
* Moderate or severe valvular disease
* Acute myocarditis
* Refractory hypertension
* Participating in other studies of drug intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with antineoplastic agents
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
At least a 10% decrease in the global longitudinal strain | 6 months
  The primary endpoint is at least a 10% decrease in the global longitudinal strain, determined using cardiac 2D STE and compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Cui, Doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Zhenyu Tian, Beijing, China

IPD SHARING:
Plan to Share IPD: No